CLINICAL TRIAL: NCT05950334
Title: A Phase 1 Study of FT522 in Combination With Rituximab in Participants With Relapsed/Refractory B-Cell Lymphoma
Brief Title: FT522 With Rituximab in Relapsed/Refractory B-Cell Lymphoma (FT522-101)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT522-101
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-07

CONDITIONS: Relapsed/Refractory B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab; Cyclophosphamide; fludarabine; Bendamustine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled first into a dose-escalation stage, followed by a dose optimization stage, and a dose-expansion stage.
Masking Description: The initial dose escalation stage of the study is nonrandomized; the dose optimization stage is randomized; the dose expansion stage is nonrandomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A (Experimental): Participants receive FT522 in combination with rituximab (or a rituximab biosimilar approved by a local health authority) with chemotherapy.
  Interventions: Drug: FT522; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine
- Regimen B (Experimental): Participants receive FT522 in combination with rituximab (or a rituximab biosimilar approved by a local health authority) without chemotherapy.
  Interventions: Drug: FT522; Drug: Rituximab

INTERVENTIONS:
Drug: FT522 — FT522 drug product is administered as an intravenous infusion on Days 1, 4 and 8 of a treatment cycle.
Drug: Rituximab — Rituximab will be administered as an IV infusion on Day -4 of the treatment cycle.
  Other Names: RITUXAN; TRUXIMA; RUXIENCE; RIABNI
Drug: Cyclophosphamide — Cyclophosphamide will be administered as an IV infusion at a dose of 500 mg/m^2 on Day -5, Day -4, and Day -3 of the treatment cycle.
  Arms: Regimen A
Drug: Fludarabine — Fludarabine will be administered as an IV infusion at a dose of 30 mg/m^2 on Day -5, Day -4, and Day -3 of the treatment cycle.
  Arms: Regimen A
Drug: Bendamustine — Bendamustine will be administered as an IV infusion at a dose of 90 mg/m^2 on Day -5 and Day -4 of the treatment cycle. Bendamustine may be administered as an alternative to cyclophosphamide/fludarabine.
  Arms: Regimen A

SUMMARY:
This is a phase 1 study of FT522 administered with rituximab in participants with relapsed/refractory B-cell lymphoma (R/R BCL). The primary objectives of the study are to evaluate the safety and tolerability of FT522 in combination with rituximab, and to determine the recommended phase 2 dose (RP2D) of FT522 in combination with rituximab; each objective will be assessed with or without conditioning chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B-cell lymphoma (BCL) as: (1) histologically documented lymphomas expected to express CD19 and CD20, including Grades 1 to 3B follicular lymphoma (FL), marginal zone lymphoma (MZL), Waldenstrom macroglobulinemia (WM), mantle cell lymphoma (MCL), transformed indolent non-Hodgkin lymphoma (tNHL), diffuse large B-cell lymphoma (DLBCL) [not otherwise specified], high-grade BCL, primary mediastinal BCL, and Richter transformation (RT; expansion part of study only); (2) R/R disease following at least 1 prior systemic regimen containing an anti-CD20 monoclonal antibody (mAb) for which the participant has no available curative treatment options; and (3) evaluable F-fluorodeoxyglucose (FDG)-avid disease, or measurable disease defined by at least one bi dimensionally measurable lesion
* Male participants and female participants of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≥2
* Body weight <50 kg
* Evidence of insufficient organ function
* Receipt of any biological therapy, chemotherapy (except for rituximab), or any investigational therapy within 2 weeks prior to Day 1 or five half-lives, whichever is shorter; or localized radiation therapy to a target lesion within 14 days prior to Day 1
* Currently receiving or likely to require systemic immunosuppressive therapy, e.g., prednisone >5 mg daily, for any reason from Day -5 to Day 29, with the exception of corticosteroids as a pre medication required for conditioning chemotherapy or rituximab
* Prior allogeneic hematopoietic stem cell transplant (HSCT) or allogeneic chimeric antigen receptor (CAR) T-cell therapy within 6 months of Day 1, or ongoing requirement for systemic graft-versus-host disease (GvHD) therapy
* Receipt of an allograft organ transplant
* Non-malignant central nervous system (CNS) disease such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease or receipt of medications for these conditions in the 2-year period leading up to study enrollment
* Clinically significant cardiovascular disease
* Clinically significant infections
* Receipt of a live vaccine <6 weeks prior to start of study intervention
* Known allergy to human albumin or DMSO
* Any medical condition or clinical laboratory abnormality that per investigator or medical monitor judgement, precludes safe participation in and completion of the study, or that could affect compliance with protocol conduct or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) | From Day 1 through Day 29 of Cycle 1
  The number of participants experiencing ≥1 DLT will be reported.
Severity of DLTs | From Day 1 through Day 29 of Cycle 1
  The severity of DLTs will be determined according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE, v5.0).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 24 months
  Participants will be classified into the following tumor response categories: complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or not evaluable (NE) according to the Lugano 2014 criteria. The best overall response (BOR) will be summarized for the efficacy evaluable population. ORR is defined as the percentage of participants who achieve a PR or better during the study prior to any subsequent off-protocol anti-cancer therapy.
Duration of Response (DOR) | Up to approximately 18 months
  The DOR is defined as the time from first objective response to disease progression or death from any cause.
Duration of Complete Response (DOCR) | Up to approximately 18 months
  The DOCR is defined as the time from first CR to disease progression or death from any cause.
Progression-Free Survival (PFS) | Up to approximately 18 months
  PFS is defined as the time from first study intervention to progressive disease or death from any cause.
Overall Survival (OS) | Up to approximately 18 months
  OS is defined as the time from first dose of study intervention to death from any cause.
Area Under the Plasma-Concentration Time Curve (AUC) of FT522 | Cycle 1, Up to Day 29
  The plasma AUC of FT522 will be reported.
Maximum Plasma Concentration (Cmax) of FT522 | Cycle 1, Up to Day 29
  The plasma Cmax of FT522 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Fate Therapeutics
Locations (7):
- United States (7):
  - Advent Health, Orlando, Florida
  - Karmanos Cancer Center, Detroit, Michigan
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Tennessee Oncology, Nashville, Tennessee
  - Baylor Houston Methodist Hospital, Houston, Texas